CLINICAL TRIAL: NCT03347240
Title: Comparative Study Between the Functional Outcomes of Neuromodulation and Neuroablation Techniques for Treatment of Secondary Dystonia
Brief Title: Neuroablation Versus Neuromodulation Techniques for Treatment of Secondary Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Nada, Fellow, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4996
Record Dates: First submitted 2017-11-12; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Secondary Dystonia
MeSH Terms: conditions — Dystonic Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brain lesioning group (Active Comparator): Stereotactic lesioning of the thalamus or gloves pallidus
  Interventions: Procedure: Brain Lesioning
- Combined rhizotomy group (Active Comparator): Combined anterior and posterior lumbosacral rhizotomy
  Interventions: Procedure: Combined anterior and posterior lumbosacral rhizotomy
- Deep brain stimulation group (Active Comparator): Bilateral globus pallidus internus deep brain stimulation
  Interventions: Device: Deep brain stimulation
- Intra-thecal Baclofen infusion therapy (Active Comparator): Intra-thecal infusion pump
  Interventions: Device: Intra-thecal baclofen infusion

INTERVENTIONS:
Procedure: Brain Lesioning — Stereotactic radiofrequency lesioning of the pallidum or thalamus
  Arms: Brain lesioning group
Procedure: Combined anterior and posterior lumbosacral rhizotomy — Combined anterior and posterior lumbosacral rhizotomy
  Arms: Combined rhizotomy group
Device: Deep brain stimulation — Bilateral DBS
  Other Names: DBS
  Arms: Deep brain stimulation group
Device: Intra-thecal baclofen infusion — Intra-thecal Baclofen infusion
  Other Names: ITB
  Arms: Intra-thecal Baclofen infusion therapy

SUMMARY:
The disability inflected by dystonia encouraged the development of many neurosurgical procedures.

This is a prospective study included 120 patients suffering from intractable secondary dystonia.

They were subjected to different neurosurgical treatments and were assessed through the follow up period

DETAILED DESCRIPTION:
Background:

Secondary dystonia are the syndromes that have dystonic symptoms due to brain insult which can be associated with neonatal encephalopathy syndromes, trauma, vascular injury, infections, demyelinations, or hereditary disorders associated with neurodegenerative process. The disability inflected by dystonia encouraged the development of many neurosurgical procedures in order to improve the quality of life of these patients.

The aim of this study was to compare the outcomes of different Neuroablative and modulation techniques in treatment of secondary dystonia.

Patients and methods This is a prospective study included 120 patients suffering from intractable secondary dystonia. Ablative techniques included the brain lesioning procedure and combined anterior and posterior lumbar rhizotomy (CAPR). Modulation techniques included deep brain stimulation (DBS) and intrathecal baclofen therapy (ITB). Patients with focal dystonia were included in the Botulinum toxin injection group. Patients with generalized dystonia were included in either of the brain lesioning or the deep brain stimulation, and patients with predominant affection of both lower limbs were included in either of the (CAPR) or the (ITB) groups.

Assessment measures included the evaluation of the muscle tone, range of motion, and the Burke-Fahn-Marsden dystonia rating scale through a follow up period of one year.

ELIGIBILITY:
Inclusion Criteria:

* secondary dystonia of previous etiologies

Exclusion Criteria:

* patients who are not candidate for anaesthesia

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Burke-Fahn-Marsden dystonia rating scale | 1 year
  Dystonia rating scale Higher scores means a worse condition of the disease, while low scores indicate a less involvement of the body

SECONDARY OUTCOMES:
Modified Ashworth scale | 1 year
  Muscle tone scale
Barthel index | 1 year
  Disability score

CONTACTS AND LOCATIONS:
Overall Officials: Walid A Abdel Ghany, MD, Study Director — Associate professor

IPD SHARING:
Plan to Share IPD: No